CLINICAL TRIAL: NCT03573102
Title: Effect of SGLT2 Inhibitor on Proteinuria in Diabetic Patients
Brief Title: Effect of Sodium Glucose co Transporter 2 Inhibitor ( SGLT2) on Proteinuria in Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nahla H Tohami (Other)
Responsible Party: Sponsor-Investigator, Nahla H Tohami, Assistent lecturer of nephrology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGLT2 antiproteinuric effect
Record Dates: First submitted 2018-03-12; First posted 2018-06-29 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Nephropathies
Keywords: proteinuria , SGLT2 inhibitors , diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors; Angiotensin-Converting Enzyme Inhibitors; Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control (Active Comparator): ACE inhibitor , aspirin , statins will be given once daily
  Interventions: Drug: ACE inhibitor
- cases (Experimental): SGLT2 inhibitors will be given with classic antiproteinuric drugs
  Interventions: Drug: SGLT2 inhibitor; Drug: ACE inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGLT2 inhibitor 10 mg/day
  Other Names: ACE Inhibitor
  Arms: cases
Drug: ACE inhibitor — ACE inhibitor once daily
  Other Names: Aspirin , statins

SUMMARY:
Diabetes Mellitus is the leading cause of end stage renal disease. As proven by many studies , controlling proteinuria can delay the progression to end stage renal disease.This work will study the effect of sodium glucose co transporter 2 inhibitor , a new antihyperglycemic drug , on proteinuria and to compare its effect with the effect of classic antiproteinuric drugs as angiotensin converting enzyme inhibitor , aspirin and statins.

DETAILED DESCRIPTION:
Diabetic nephropathy involves progressive stages including glomerular hyperfilteration , microalbuminuria , overt proteinuria and a decline in glomerular filteration rate leading to end stage renal disease.

Despite all the available interventions available for diabetic patients including tight glycemic control , and blood pressure control , using angiotensin converting enzyme inhibitors, angiotensin II receptor antagonist renal disease remains prevalent and progress in these patients.

The newer therapy of diabetes is the use of sodium glucose cotransporter 2 inhibitor as it has the potential of renoprotection in patients with diabetic nephropathy just as ACEI and ARBS to reduce glomerular hyperfilteration .This action may reduce albuminuria.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with type 2 diabetes.
* controlled diabetes.
* patients with proteinuria

Exclusion Criteria:

* patients with proteinuria due to other disease.
* patients with HbA1c >8%.
* patients with uncontrolled hypertension.
* patients with chronic liver disease.
* patients with type 1 diabetes .
* patients already on the same drug ( dapagliflozine).
* patients with raised serum creatinine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
decrease in proteinuria | 6 months
  improvement of proteinuria in patients receiving dapagliflozine

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Sharkawy, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lotfy M, Adeghate J, Kalasz H, Singh J, Adeghate E. Chronic Complications of Diabetes Mellitus: A Mini Review. Curr Diabetes Rev. 2017;13(1):3-10. doi: 10.2174/1573399812666151016101622. PMID 26472574